CLINICAL TRIAL: NCT06411262
Title: Pilot Study Investigating Intensity and Quality of Movement Performed During a Parkiboks Session
Acronym: Parkiboks
Status: Recruiting | Type: Observational
Sponsor: Hasselt University (Other)
Responsible Party: Principal Investigator, Peter Feys, Professor Peter Feys, Hasselt University
Other Study IDs: CME2024/009
Record Dates: First submitted 2024-05-08; First posted 2024-05-13 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Parkiboks — A non-contact boxing sessions for individuals with Parkinson disease, made-up of 3 sections: a warm-up, a boxing section, a cool-down. Each section is split into a range of exercises. The session is led by a boxing coach with training and expertise in Parkinson disease.

SUMMARY:
Studies have shown that non-contact boxing benefits individuals with Parkinson disease. Yet, the content of such sessions, has not yet been investigated. The following research question has therefore been asked: What is the physical intensity, in terms of both movement quality and quantity, as well as cardiovascular demand, in a group of individuals with Parkinson's disease during a one-hour session of Parkiboks? Though the study is exploratory, the investigators hypothesize to observe increases in cardiovascular activity during the session, as well as a high number of upper-limb repetitions of near maximal range of motion.

ELIGIBILITY:
Inclusion Criteria:

* Official diagnosis of Parkinson disease Active participants of a non-contact boxing group for people with Parkinson disease located in Turnhout, Belgium Participating in non-contact boxing sessions for at least one month prior to the study

Exclusion Criteria:

* Unable to read and understand the informed consent document Individuals who are wheelchair-bound

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All individuals with Parkinson disease who have been active participants of the non-contact boxing sports group in Turnhout, Beligum, will be invited to participate.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2024-05-08 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Upper-limb kinematics | Measured during one complete non-contact boxing session, which lasts one hour.
  Movella DOT sensors secured on the left and right wrists.
Cardiovascular load | Measured during one complete non-contact boxing session, which lasts one hour.
  Polar heart rate sensor secured by a strap around the thorax.

SECONDARY OUTCOMES:
Motor impairments | Filled in at the beginning of the session, together with the examinator.
  Score obtained on the Hoehn and Yahr scale. Scores range from 0 to 5, where 0 represents no physical impairments and 5 represents worse impairments.
Activity limitations related to motor impairments | Filled in by the participant prior to the session.
  Score obtained on the Movement Disorder Society-Unified Parkinson's Disease Rating Scale (PDS-UPDRS) Part II (Motor experiences of daily living). Scores range from 0 to 52, where 0 indicates no activity limitations related to motor impairments and 52 indicates worse limitations.
Fatigue severity | Filled in by the participant prior to the session.
  Score obtained on the Fatigue Severity scale. Scores range from 1 to 7, where 1 represents no fatigue and 7 indicates high severity of fatigue.
Fear of falling | Filled in by the participant prior to the session.
  Score obtained on the Falls Efficacy scale - International. Scores range from 16 to 64, where 16 represent no fear of falling, and 64 represents worse fear of falling.
Perceived exertion during the completed session | Filled in by the participant at the end of the session.
  Score obtained on the Borg'scale for rating perceived exertion. Scores range from 6 to 20, where 6 presents no perceived exertion, and 20 represents maximal perceived exertion.
Perceived balance difficulty during the session | Filled in by the participant at the end of the session.
  Score obtained on a visual analogue scale. Scores from 0 to 10, where 0 represents no difficulty with balance during the session, and 10 represent highest level of difficult with balance during the session.

OTHER OUTCOMES:
Demographic parameters | Filled in by the participant prior to the session.
  Self-reported questionnaire related to age, gender, height, weight, sports participation, comorbidities, year of diagnosis of Parkinson and dopamine supplementation.
Most challenging exercise | Filled in by the participant at the end of the session.
  Self-reported account of the exercise the participant found to be most challenging during the session.
Most tiring exercise | Filled in by the participant at the end of the session.
  Self-reported account of the exercise the participant found to be most tiring during the session.

CONTACTS AND LOCATIONS:
Locations (1):
- UHasselt, Diepenbeek, Flanders, Belgium

IPD SHARING:
Plan to Share IPD: Undecided